CLINICAL TRIAL: NCT03641482
Title: Effect of NBF Gingival Gel Application in Controlling Post-surgical Complications After Impacted Lower Third Molar Surgery
Brief Title: NBF Gingival Gel Application After Impacted Lower Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Bio Nature Essences S.L (Unknown)
Responsible Party: Principal Investigator, Rosa María López-Pintor Muñoz, Associate professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0002
Record Dates: First submitted 2018-08-01; First posted 2018-08-22 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Alveolar Osteitis
Keywords: third molar surgery; oral surgery; propolis; NBF gingival gel; post-surgical complications; clinica trial
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: split mouth design
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NBF (Active Comparator): Propolis Extract, Ascorbic Acid, Tocopherol Acetate, Sodium-Monofluorophosphate, Silicon Dioxide, Glycerin, D-sorbitol, Polyethyleneglycol 150, Sodium Carboxymethylcellulose, Xylitol, Sterol Glycoside, Peppermint Oil, L-Menthol, Methyl Hydroxybenzoate and Deionized Water
  Interventions: Drug: NBF
- Placebo (Placebo Comparator): Sodium-Monofluorophosphate, Silicon Dioxide, Glycerin, D-sorbitol, Polyethyleneglycol 150, Sodium Carboxymethylcellulose, Xylitol, Sterol Glycoside, Peppermint Oil, L-Menthol, Methyl Hydroxybenzoate and Deionized Water
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: NBF — Once the molar is extracted, the socket is cleaned with water, NBF gel is introduced, and the flap is closed. Then, the patients are instructed to apply NBF Gel in the surgical wound 3 times per day for 7 days after brushing their teeth. Previously they have to dry the area of the wound with gauze.
  Arms: NBF
Device: Placebo — Once the molar is extracted, the socket is cleaned with water, placebo gel is introduced, and the flap is closed. Then, the patients are instructed to apply placebo gel in the surgical wound 3 times per day for 7 days after brushing their teeth. Previously they have to dry the area of the wound with gauze.
  Arms: Placebo

SUMMARY:
Background: Alveolar osteitis is one of the most frequent complications after lower third molar extraction, and is usually accompanied by inflammation, pain and poor wound healing. Several local interventions have been used to reduce these complications with limited effectiveness.

Purpose: To clinically evaluate the use of propolis extract, nanovitamin C and nanovitamin E gel for the prevention of surgical complications related to impacted lower third molar extraction.

Methods: A randomized, triple-blind, split-mouth, pilot study is being performed in patients needing bilateral lower third molar extraction with similar surgical difficulty. Surgical extractions are randomly being performed and NBF gingival gel (TG) or placebo (PBG) are randomly being applied inside postextraction sockets by a blinded surgeon. The patients are being instructed to apply it 3 times/day in the surgical wound for 7 days. One month later, the contralateral wisdom tooth is being extracted and the opposite gel is being applied. Alveolar osteitis (AO) is being diagnosed following Blum's criteria. Swelling is being assessed by measuring the facial perimeter. Wound healing is being evaluated with a semi-quantitative scale as good, satisfactory or insufficient. Postoperative pain is being recorded using a visual analog scale (VAS) for 7 days. Analgesic pill intake is being recorded by each patient. Variables are being registered by a blinded researcher to 3M extractions at one, two, three and seven postoperative days.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are:

* cooperative adult patients able to fulfil the study protocol,
* needing surgical extractions of both lower third molars,
* with similar surgical difficulty according to Pederson scale.

Exclusion Criteria:

The exclusion criteria are

* refuse to participate in the study,
* failure to attend 24, 48, and 72 hours, as well as, 7 days post-surgical appointment visits,
* smokers,
* systemic diseases as diabetes mellitus or being immunosuppressed,
* patients who take local or systemic antibiotics less than 3 months ago, anti-inflammatory or anticoagulant medication in the previous 4 weeks,
* patients who require antibiotic prophylaxis,
* pregnant or breastfeeding women,
* patients with chronic periodontitis in active phase or
* with history of allergies to any of the components of local anaesthetics, antibiotics, AINEs, or NBF gingival gel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Alveolar Osteitis: intense neuralgic pain in the post-extraction socket in the second or third postoperative day that do not disappear with analgesics beside a partially or totally disintegrated clot | from baseline to 24, 48, 72 hours post intervention
  yes or no

SECONDARY OUTCOMES:
Swelling: it was evaluated with a flexible metric tape measuring the facial perimeter from trago to pogonion. A first measurement was made before surgery, which was compared with the measurements taken at 24, 48 and 72 hours of the extraction. | from baseline to 24, 48, 72 hours and 7 days post intervention
  changes
Trismus: it was assessed measuring the maximum opening from the inter incisive points. | from baseline to 24, 48, 72 hours and 7 days post intervention
  changes
Wound healing: it was assessed with a semi-quantitative scale (good, satisfactory or insufficient). | from baseline to 1 week post intervention
  changes
Post extraction pain: it was recorded using a visual analog scale, ranging from 0 (no pain) to 10 (the worst pain imaginable) at 9 pm of 7 consecutive days. | from baseline to 1 week post intervention
  changes
Number of rescue analgesic pills consumption: recorded for the first 3 days by the patients. | from baseline to 3 days post intervention
  number

REFERENCES:
- [Background] Blum IR. Contemporary views on dry socket (alveolar osteitis): a clinical appraisal of standardization, aetiopathogenesis and management: a critical review. Int J Oral Maxillofac Surg. 2002 Jun;31(3):309-17. doi: 10.1054/ijom.2002.0263. PMID 12190139
- [Background] Haraji A, Rakhshan V, Khamverdi N, Alishahi HK. Effects of intra-alveolar placement of 0.2% chlorhexidine bioadhesive gel on dry socket incidence and postsurgical pain: a double-blind split-mouth randomized controlled clinical trial. J Orofac Pain. 2013 Summer;27(3):256-62. doi: 10.11607/jop.1142. PMID 23882458
- [Background] Madrazo-Jimenez M, Rodriguez-Caballero A, Serrera-Figallo MA, Garrido-Serrano R, Gutierrez-Corrales A, Gutierrez-Perez JL, Torres-Lagares D. The effects of a topical gel containing chitosan, 0,2% chlorhexidine, allantoin and despanthenol on the wound healing process subsequent to impacted lower third molar extraction. Med Oral Patol Oral Cir Bucal. 2016 Nov 1;21(6):e696-e702. doi: 10.4317/medoral.21281. PMID 27475700